CLINICAL TRIAL: NCT06502704
Title: Bile Acids and Microbiome - Possible Novel Progression Factors and Diagnostic Indicators in Early Colorectal Carcinogenesis
Brief Title: Bile Acids and Microbiome in Early Colorectal Carcinogenesis
Status: Recruiting | Type: Observational
Sponsor: Vilnius University (Other)
Collaborators: Vilnius University Hospital Santaros Klinikos (Other)
Responsible Party: Sponsor
Other Study IDs: 2024/5-1587-1047
Record Dates: First submitted 2024-06-17; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Colorectal Neoplasms; Colorectal Cancer; Colorectal Polyp; Microbiome; Bile Acid Malabsorption
Keywords: Colorectal Neoplasms; Colorectal Cancer; Colorectal Polyp; Microbiome; Bile Acid
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fecal, Blood, Urine and gut biopsy samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control: No pathology upon colonoscopy
- Small adenoma: < 1cm size polyp upon colonoscopy
- Large adenoma: > 1cm size polyp upon colonoscopy
- Cancer: Adenocarcinoma upon colonoscopy

SUMMARY:
Currently colorectal cancer pathogenesis is mainly explained by the adenoma-carcinoma sequence theory that was proposed more than half a century ago. It mainly focuses on the explanation of genetic mutations that develop throughout the disease course. However, several studies argue that there are also noticeable bile acid metabolism changes and microbiome composition changes within in colorectal cancer patients. However, carcinoma is the final step in the sequence, and prior steps are noticeably less well studied. Thus, the investigators hypothesize, that changes within microbiome and the changes in the urine, serum and gut bile acid composition further leads to the development of colorectal adenoma and subsequent invasive carcinoma.

Adult participants (15 per group) referred for colonoscopy and histologically diagnosed with small (<1cm) adenomas, large (>1cm) adenomas, invasive CRC will be included in the study, as well as 15 healthy controls. Fecal samples will be collected from all participants before bowel preparation. Additionally, urine and serum samples will be collected. Participants will undergo polypectomy, endoscopic mucosal resections, depending on the location, size and histology of the polyp found. During colonoscopy the mucosal biopsy specimens from the lesion and from the healthy bowel -terminal ileum, and colon will be obtained using sterile biopsy forceps. The collected samples will be stored for bile acid and microbiome analysis and for possible further pathology and genetic testing. Healthy participants without visible colorectum pathology during colonoscopy will undergo colon and terminal ileum mucosal sampling.

The investigators plan to evaluate the correlation between the urine and gut microbiome changes and bile acid composition and concentration in adenoma-carcinoma sequence and possibly determine novel bile acids. In addition, fecal, urine and tissue samples will be explored for gut microbiota and bile acid composition changes in healthy and along the adenoma-carcinoma sequence, with the possibility to propose a diagnostic test.

ELIGIBILITY:
Inclusion Criteria:

- Patients that have clinical indications for colonoscopy

Exclusion Criteria:

* Pregnancy
* Immunocompromised
* Previously diagnosed colorectal diseases
* Radiotherapy to the pelvis
* Long term antibiotic use within 6 months
* Continuous use of proton pump inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: > 18 years of age, atients that have clinical indications for colonoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-07-05 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Microbiome and bile acid composition correlation to dysplastic changes | Through study completion, an average of 2 years
  Microbiome and bile acid composition changes will be detected and correlated with progression of the dysplastic changes within the epithelium of the large bowel.

SECONDARY OUTCOMES:
Bile acid composition in healthy participants | Through study completion, an average of 2 years
  Compare bile acid composition of healthy controls to patients with early and advanced adenomas and colorectal cancer, novel bile acid identification that could play a role in the adenoma-carcinoma sequence and identify the diagnostic potential of bile acid composition patterns
Bile acid composition in urine, stool and serum | Through study completion, an average of 2 years
  Determine the bile acid composition in urine, stool and serum of healthy controls

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Poskus, PhD, Principal Investigator — Vilnius University
Locations (1):
- Vilnius University Hospital Santaros Klinikos, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: No